CLINICAL TRIAL: NCT05949996
Title: Evaluation of a Program for Routine Implementation of Symptom Distress Screening and Referral in Cancer Care: a Stepped Wedge Cluster Randomized Trial
Brief Title: Evaluation of a Program for Routine Implementation of Symptom Distress Screening and Referral in Cancer Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Health and Medical Research Fund (Other Government)
Responsible Party: Principal Investigator, Wendy Wing Tak Lam, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: UW22-645
Record Dates: First submitted 2023-06-05; First posted 2023-07-18 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Neoplasms
Keywords: Implementation study; Symptom distress screening; Survivorship care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This study will use a stepped wedge cluster randomized controlled trial design in which the intervention is introduced stepwise across study units. All study units will be asked to sign a consent form for study participation and will start with the 4-month control situation (i.e. No nurse-led symptom distress screening program at the beginning of the study). Then, the study units are randomized to one of the three roll-out schedules with a 4-month duration each. At each time point, a new group of 2 or 3 study units will cross over from the control condition to the implementation condition. For each eligible patient who is approached and being screened for symptom distress, the HA nursing staff will explain the objective of the symptom distress screening and obtain written consent for agreeing to participate in the screening program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implementation condition (Experimental): Under implementation condition, a nurse-led symptom distress screening program will be implemented using 5 implementation strategies including training, audit and feedback, facilitation and adaptable workflow.
  Interventions: Other: A nurse-led symptom distress screening program
- Control condition (No Intervention): The control condition is the usual clinical outpatient operation without the specific implementation program (i.e. applying the five implementation strategies including training, audit and feedback, facilitation and adaptable workflow) for standardized routine symptom distress screening. Prior to the start of the first 4-month control condition, we will meet each study unit and brief the staff about the purpose of this implementation study, as well as the introduction of the symptom distress screening tool. The symptom distress screening tool and referral forms will be given to the study sites. The staff are encouraged to screened and referred all eligible patients to JCICC, a local cancer care centre. In contrast to the intervention condition, there will be no half-day skill training workshop and no weekly audit and feedback report delivered and discussed with the site facilitator. We will keep the recording of the briefing session for fidelity assessment.

INTERVENTIONS:
Other: A nurse-led symptom distress screening program — Five implementation strategies will be conducted individually for each of the study unit at the timepoint when the study unit is being randomly allocated to the implementation condition. For each study unit, all nurses will first receive a half-day training. Each study unit under the implementation condition will receive weekly audit and feedback reports to summarize the proportion of eligible patients, proportion of eligible patients being screened, proportion of patients appropriately referred to JCICC. The senior research assistant with a nursing background will receive training and mentoring from the PI and will be the guided facilitator. The guided facilitator will conduct weekly site visits to address operational issues arise during the implementation. Lastly, while the choice of symptom assessment tool and referral criteria are standardized and cannot be modified, the routine workflow for each study unit can be adjusted according to its context and resources.
  Arms: Implementation condition

SUMMARY:
This study proposes to evaluate the process and outcome of an implementation program designed to implement nurse-led symptom distress screening and referral into routine cancer care clinics. Specifically, using a stepped-wedge cluster randomized controlled trial, This study aim to test if a systematic symptom distress screening program increases the proportion of eligible patients screened and referred compared to usual control. For process evaluation, this study will use qualitative methods to assess the experience and response to the implementation program.

DETAILED DESCRIPTION:
This study proposes to evaluate the process and outcome of an implementation program designed to implement nurse-led symptom distress screening and referral into routine cancer care clinics. Specifically, using a stepped-wedge cluster randomized controlled trial, this study aim to test if a systematic symptom distress screening program (i.e. using the five implementation strategies including training, audit, feedback, facilitation and adaptable workflow) increases the proportion of eligible patients screened and referred compared to usual control under which no implementation strategies will be used to facilitate the adoption of the systematic symptom distress screening and referral. The investigator hypothesize that (1) the intervention will increase the proportion of eligible patients screened; (2) the intervention will increase the proportion of patients with moderate to severe symptom distress referred for psychosocial support.

For process evaluation, this study will use qualitative methods to assess the experience and response to the implementation program.

ELIGIBILITY:
Inclusion Criteria:

* All cancer patients within two years post-treatment attending the specialized outpatient clinics for surveillance will be eligible for symptom distress screening, with no exclusions by any demographic and clinical characteristics.

Exclusion Criteria:

* All cancer patients beyond two years post-treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2772 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in the number of eligible patient screened | Pre- and post-implementation phase, up to 24 months
  The primary outcome (the measurement of the reach) is the changes in the number of eligible patients screened. Using a standardized reporting form, each study site will be asked to submit a weekly record of a total number of eligible patients per clinic and the number of patients screened.
Change in the number of eligible patient referred | Pre- and post-implementation phase, up to 24 months
  The primary outcome (the measurement of the reach) is the changes in the number of eligible patients referred based on the predefined scores. Using a standardized reporting form, each study site will be asked to submit a weekly record of a total number of eligible patients per clinic and the number of patients referred.

SECONDARY OUTCOMES:
Change in referral uptake | Pre- and post-implementation phase, up to 24 months
  The secondary outcome is the change in uptake of the referral, i.e. the proportion of referred patients accepting services.
Process evaluation in providers by conducting qualitative interviews | post-implementation phase, up to 24 months
  Using qualitative approach with service providers (i.e. the nurses) to identify facilitators and barriers for the implementation of the symptom distress screening program, as well as their overall experience. All nursing staff from the study units involved in the symptom distress screening will be invited to join the qualitative study at the post-implementation phase.
Process evaluation in patients by conducting qualitative interviews | post-implementation phase, up to 24 months
  We will also conduct qualitative interviews to explore patients' experiences with symptom distress screening and referral if appropriate. Patients who are referred for support services will be approached by the research assistant who will explain the purpose of the study and nature of participation, with an emphasis on confidentiality and anonymity. If agreeing to participate, the RA will obtain a written consent and each subject will subsequently participate in in-depth interview by a trained interviewer. For patients who decline to be referred for support services, we will ask the nursing staff to invite the patients to join the qualitative study. We will recruit patients from both implementation and control conditions as it will enable us to compare patients' experienc.
Number of staff receiving training | pre-implementation phase, up to 24 months
  All nurses will first receive a half-day training on how to administer the symptom distress screening tool, evaluate patients' reported symptom distress, refer patients to and follow-up for referred patients. We will record the number of invited staff attending the half-day training workshop.
Change in staff knowledge about the implementation of the screening programme assessed using categorical Likert scales | pre- and post-training workshop, and post-implementation phase, up to 24 months
  We will assess the staff knowledge at pre- and post-training workshop and again at the end of the implementation study using a 6 points-categorical Likert scale (0-5) for participants' knowledge about the implementation of the screening program. Such information will be served as implementation indicators to facilitate the interpretation of the study findings.
Change in staff's belief in the symptom distress screening programme assessed using categorical Likert scales | pre- and post-training workshop, and post-implementation phase, up to 24 months
  We will assess the staff's belief at pre- and post-training workshop and again at the end of the implementation study using a 6 points-categorical Likert scale (0-5) for participants' beliefs towards the symptom distress screening programme. Such information will be served as implementation indicators to facilitate the interpretation of the study findings.
Change in staff self-efficacy in administrating the symptom distress screening programme assessed using categorical Likert scales | pre- and post-training workshop, and post-implementation phase, up to 24 months
  We will assess the staff's self-efficacy at pre- and post-training workshop and again at the end of the implementation study using a 6 points-categorical Likert scale (0-5). Such information will be served as implementation indicators to facilitate the interpretation of the study findings.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Wing Tak Lam, PhD, Principal Investigator — School of Public Health, The University of Hong Kong
Locations (10):
- Hong Kong (10):
  - JCICC, Hong Kong
  - Kwong Wah Hospital-Breast Center, Hong Kong
  - North District Hospital, Hong Kong
  - Pamela Youde Nethersole Eastern Hospital-Department of oncology, Hong Kong
  - Prince of Wales Hospital-Department of Surgery, Hong Kong
  - Queen Mary Hospital-Department of Obstetrics & Gynaecology, Hong Kong
  - Queen Mary Hospital-Department of Oncology, Hong Kong
  - Queen Mary Hospital-Department of Surgery, Hong Kong
  - The University of Hong Kong Jockey Club Institute of Cancer Care, Hong Kong
  - Tung Wah Hospital-Department of Surgery, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available from the PI upon reasonable request.
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication
Access Criteria: Information will be available from the PI upon reasonable request. The author to review requests is the PI.

REFERENCES:
- See also: HKU JCICC, a local cancer care centre — https://jcicc.med.hku.hk/?lang=en